CLINICAL TRIAL: NCT04559256
Title: Transcatheter Tricuspid Valve Interventions and Right Ventricular Function: Evaluation with Cardiopulmonary Exercise Testing
Brief Title: Tricuspid Cardiopulmonary Exercise Study
Acronym: TRCPET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Principal Investigator, Muhammed Gerçek, Principal Investigator, Heart and Diabetes Center North-Rhine Westfalia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDZ-KA_018_MG
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Tricuspid Regurgitation
Keywords: Tricuspid Regurgitation; Cardiopulmonary Exercise Testing
MeSH Terms: conditions — Tricuspid Valve Insufficiency | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tricuspid Cardiopulmonary Exercise testing (Other): Patient receiving cardiopulmonary exercise testing
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary Exercise Testing — Patients will receive a cardiopulmonary exercise testing before and 3-month after tricuspid intervention

SUMMARY:
Tricuspid regurgitation (TR), which in close to 90% of cases is functional as a consequence of left-sided heart failure, left heart valve abnormalities or pulmonary (vascular) disease, is associated with adverse patient outcomes . Due to the increased risk of surgical tricuspid valve repair or replacement compared to surgery in left-sided valve disease TR is often undertreated. Treatment options for the tricuspid valve have so far been limited. Conservative therapy over longer. periods usually results in refractoriness to diuretic treatment. Surgical therapy is associated with a high rate of in-hospital mortality (8.8%), the cause of which is not yet fully understood but may partly be explained by the hemodynamic challenge that cardiopulmonary bypass imposes on the often already-dysfunctional right ventricle. Recently, transcatheter strategies have been developed and have shown promising results. Despite the promising data it has so far not be determined objectively whether interventional treatment of isolated tricuspid regurgitation improves exercise capacity and what role right ventricular function plays in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Chronic tricuspid regurgitation 2+ to 4+ on a scale of 4+ (moderate to severe) with annular diameter ≥ 40 mm with valve systolic pulmonary pressure (sPAP) ≤ 60 mmHg
* New York Heart Association (NYHA) Class II-IV
* Symptomatic despite Guideline Directed Medical Therapy (GDMT); at minimum patient on diuretic regimen
* Left ventricular ejection fraction ≥ 30%
* Symptomatic despite Guideline Directed Medical Therapy (GDMT); at minimum patient on diuretic regimen
* The local site Heart Team concur that surgery will not be offered as a treatment option
* Written informed consent in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Inability to perform cardiopulmonary exercise test
* Aortic, mitral and/or pulmonic valve stenosis and/or regurgitation ≥ moderate
* Previous tricuspid valve repair or replacement
* Severe precapillary pulmonary hypertension (PVR>6 WE)
* Cerebrovascular accident (CVA) within the past 6 months
* Presence of trans-tricuspid pacemaker or defibrillator leads which cause impingement of the tricuspid valve leaflet as evaluated by echocardiography
* Subject is on chronic dialysis and/or anemia (Hb < 9 g/L)
* Myocardial infarction or known unstable angina within 30 days prior to the index procedure
* Any percutaneous coronary intervention or transcatheter valvular intervention within 30 days prior to the index procedure or planned 3 months post the index procedure
* Previous tricuspid valve repair or replacement
* Life expectancy of less than 12 months
* Patients with cardiac cachexia
* Echocardiographic evaluation not available or not suitable for analysis at baseline
* Unsuitable anatomy for transcatheter tricuspid intervention
* Key information from patients (e.g. NYHA, TR grade) not available
* Known allergy or intolerance against the studied device
* Persons held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Influence of transcatheter tricuspid intervention on peak oxygen uptake | 3 month
  Changes on maximal oxygen uptake (peak VO2) assessed by cardiopulmonary exercise testing (CPET, spiroergometry) after transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on duration of submaximal exercise tolerance | 3 month
  Changes on the duration of submaximal exercise tolerance assessed by exercise time during high-intensity constant-work rate endurance tests (CWRET) after transcatheter tricuspid intervention

SECONDARY OUTCOMES:
Influence of transcatheter tricuspid intervention on the minute ventilation/carbon dioxide production slope in the cardiopulmonary exercise testing | 3 month
  Changes on the minute ventilation/carbon dioxide production slope in the cardiopulmonary exercise testing after transcatheter tricuspid intervention
Prevalence of oscillatory respiration pattern | 3 month
  Detection of oscillatory respiration pattern before and 3 months after transcatheter tricuspid intervention
Exercise Testing with 6 min walking test | 3 month
  Changes on walked distance after transcatheter tricuspid intervention
Prevalence of moderate to severe or severe tricuspid regurgitation | 3 month
  Detection of the prevalence of moderate to severe or severe tricuspid regurgitation after transcatheter tricuspid intervention
Rehospitalization rate for heart failure | 3 month
  Detection of rehospitalization rate after transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on NYHA class | 3 month
  Changes on NYHA class after transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on quality of life | 3 month
  Changes on the Minnesota Living with Heart Failure Questionnaire score after transcatheter tricuspid intervention (0-105 points on a global scale, with 0 points representing a very good quality of life and 105 points representing a very reduced quality of life)
Influence of transcatheter tricuspid intervention on the left an right ventricle | 3 month
  Echocardiographic assessment of left and right ventricular remodeling after transcatheter tricuspid intervention
Influence of transcatheter tricuspid intervention on serum N terminal-proBNP level | 3 month
  Changes on serum N terminal-proBNP-level after transcatheter tricuspid intervention

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Gerçek, MD, Principal Investigator — Heart and Diabetes Center North-Rhine Westfalia
Locations (1):
- Herz- und Diabeteszentrum, NRW, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No